CLINICAL TRIAL: NCT02203578
Title: A Pilot Study of Romidepsin for Therapy of Graft-versus-Host Disease
Brief Title: Romidepsin in Treating Patients With Steroid-Refractory Graft-versus-Host Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: slow accrual
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 021309; NCI-2014-01411 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 021309 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH); Pro2014004116 (Other: IRB number)
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Results first posted 2017-03-30 (Actual); Last update posted 2017-03-30 (Actual); Status verified 2017-02

CONDITIONS: Graft Versus Host Disease
MeSH Terms: conditions — Graft vs Host Disease | interventions — romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Supportive care (romidepsin) (Experimental): Patients receive romidepsin IV over 4 hours on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: romidepsin; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: romidepsin — Given IV
  Other Names: FK228; FR901228; Istodax
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This pilot clinical trial studies romidepsin in treating patients with graft-versus-host disease (GVHD) that has not responded to treatment with steroids. Romidepsin may be an effective treatment for graft-versus-host disease caused by a bone marrow or stem cell transplant.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if romidepsin should be developed as a therapy for patients with steroid-refractory GVHD.

OUTLINE:

Patients receive romidepsin intravenously (IV) over 4 hours on days 1, 8, and 15. Treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3 and 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with steroid (or immunosuppressive therapy [IST]) refractory acute GVHD (aGVHD) or chronic GVHD (cGVHD)
* Absolute neutrophil count >= 750/mm^3
* Platelet count >= 50,000/mm^3
* Corrected QT interval (QTc) =< 480 msec
* Bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x ULN
* Serum potassium >= 3.8 mmol/L
* Serum magnesium >= 1.8 mg/dL
* Serum creatinine =< 2.0 mg/dl
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-3
* Patients may undergo electrolyte repletion therapy to meet eligibility requirements
* Patients must be scheduled for tapering doses of (or no longer treated with):

  * Cyclosporine;
  * Tacrolimus;
  * Sirolimus;
  * Steroids (patients may be on physiologic doses of steroids)
* Patients receiving extracorporeal photopheresis must discontinue extracorporeal photopheresis or placed on a tapering schedule;
* Any prior therapy for GVHD must be completed and discontinued with the exception of the above;
* Patients with breakpoint cluster region (bcr)-ABL proto-oncogene 1 (abl) associated malignancies may be on a tyrosine kinase inhibitor as malignant disease therapy or prophylaxis
* There must be no uncontrolled active infections or medical conditions that the investigator feels will compromise the safety of the treatment and/or the assessment of the efficacy of therapy
* The patient must be aware of the high risk and experimental nature of the treatment and provide informed consent
* Negative serum pregnancy test at the time of enrollment for females of childbearing potential
* For males and females of child-producing potential, use of effective contraceptive methods during the study and for at least 6 months after the last dose of romidepsin

Exclusion Criteria:

* Active/uncontrolled infection
* Evidence of relapsed disease
* Life expectancy < 12 weeks
* Pregnant or breast feeding females
* Prior therapy with romidepsin
* Known seropositive for or active viral infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV); patients who are seropositive because of hepatitis B virus vaccine are eligible
* Any known cardiac abnormalities such as:

  * Congenital long QT syndrome
  * QTc interval >= 480 milliseconds;
  * Myocardial infarction within 6 months of course 1, day 1 (C1D1); subjects with a history of myocardial infarction between 6 and 12 months prior to C1D1 who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event may participate;
  * Other significant electrocardiogram (ECG) abnormalities including 2nd degree atrio-ventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min);
  * Symptomatic coronary artery disease (CAD), e.g., angina Canadian class II-IV; in any patient in whom there is doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
  * An ECG recorded at screening showing evidence of cardiac ischemia (ST depression of >= 2 mm, measured from isoelectric line to the ST segment); if in any doubt, the patient should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present;
  * Congestive heart failure (CHF) that meets New York Heart Association (NYHA) class II to IV definitions and/or ejection fraction < 40% by multi gated acquisition (MUGA) scan or < 50% by echocardiogram and/or magnetic resonance imaging (MRI);
  * A known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), Torsade de Pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD);
  * Hypertrophic cardiomegaly or restrictive cardiomyopathy from prior treatment or other cause;
  * Any cardiac arrhythmia requiring an anti-arrhythmic medication (excluding stable doses of beta-blockers)
* Uncontrolled hypertension, i.e., blood pressure (BP) of >= 160/95; patients who have a history of hypertension controlled by medication must be on a stable dose (for at least one month) and meet all other inclusion criteria; or
* Patients taking drugs leading to significant QT prolongation must have an ECG prior to each treatment
* Concomitant use of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors
* Concomitant use of medications known to induce a disulfiram-like reaction to alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-11; Primary Completion 2016-06-14 (Actual); Study Completion 2016-06-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited through the Rutgers Cancer Institute of New Jersey. The study was open to accrual on 11/20/2014 and was closed by the Principal Investigator on 6/14/2016 due to slow accrual.
Pre-assignment Details: We are reporting results on 1 eligible participant.
Period: Overall Study
Arm/Group | Supportive Care (Romidepsin)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Participants > 18 years old with steroid (or IST) refractory aGVHD or cGVHD were enrolled.
Arm/Group | Supportive Care (Romidepsin)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 49 [49 to 49]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of aGVHD
Time Frame: At 28 days after initiation of romidepsin
Population: Study was terminated early due to slow accrual and insufficient data was collected to assess this outcome measure.
Arm/Group | Supportive Care (Romidepsin)
Number analyzed (Participants) | 0
Value | 0

2. Primary Outcome: Incidence of cGVHD
Time Frame: At 1 month after initiation of romidepsin
Population: Study was terminated early due to slow accrual and insufficient data was collected to assess this outcome measure.
Arm/Group | Supportive Care (Romidepsin)
Number analyzed (Participants) | 0
Value | 0

3. Primary Outcome: Incidence of cGVHD
Time Frame: At 3 months after initiation of romidepsin
Population: Study was terminated early due to slow accrual and insufficient data was collected to assess this outcome measure.
Arm/Group | Supportive Care (Romidepsin)
Number analyzed (Participants) | 0
Value | 0

4. Primary Outcome: Incidence of cGVHD
Time Frame: At 6 months after initiation of romidepsin
Population: Study was terminated early due to slow accrual and insufficient data was collected to assess this outcome measure.
Arm/Group | Supportive Care (Romidepsin)
Number analyzed (Participants) | 0
Value | 0

5. Primary Outcome: Incidence of cGVHD
Time Frame: At 9 months after initiation of romidepsin
Population: Study was terminated early due to slow accrual and insufficient data was collected to assess this outcome measure.
Arm/Group | Supportive Care (Romidepsin)
Number analyzed (Participants) | 0
Value | 0

6. Primary Outcome: Incidence of cGVHD
Time Frame: At 12 months after initiation of romidepsin
Population: Study was terminated early due to slow accrual and insufficient data was collected to assess this outcome measure.
Arm/Group | Supportive Care (Romidepsin)
Number analyzed (Participants) | 0
Value | 0

7. Secondary Outcome: Total Duration of Immunosuppressive Therapy
Time Frame: Up to 12 months after initiation of romidepsin
Population: Study was terminated early due to slow accrual and insufficient data was collected to assess this outcome measure.
Arm/Group | Supportive Care (Romidepsin)
Number analyzed (Participants) | 0
Value | 0

8. Secondary Outcome: Rate of Documented Infection
Time Frame: Up to 12 months after initiation of romidepsin
Population: Study was terminated early due to slow accrual and insufficient data was collected to assess this outcome measure.
Arm/Group | Supportive Care (Romidepsin)
Number analyzed (Participants) | 0
Value | 0

9. Secondary Outcome: T Cell Kinetics - Reconstitution
Time Frame: Up to 12 months after initiation of romidepsin
Population: Study was terminated early due to slow accrual and insufficient data was collected to assess this outcome measure.
Arm/Group | Supportive Care (Romidepsin)
Number analyzed (Participants) | 0
Value | 0

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over 60 days.
Description: CTCAE version 4.0 was utilized.
Arm/Group | Supportive Care (Romidepsin)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Romidepsin) (N=1)
Endocarditis infective (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Supportive Care (Romidepsin) (N=1)
Nausea (Gastrointestinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes